CLINICAL TRIAL: NCT00969475
Title: The Effects of Fractional CO2 Resurfacing Prior to Complex Wound Closure
Brief Title: The Effects of Fractional Carbon Dioxide (CO2) Laser Treatment Prior to Wound Closure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Moy-Fincher Medical Group (Other)
Responsible Party: Ronald Moy, MD, Moy-Fincher Medical Group
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MF-01
Record Dates: First submitted 2009-08-29; First posted 2009-09-01 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Scars
Keywords: scar revision; intraoperative; fractional carbon dioxide laser
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Half of each subject's wound will not be treated.
- Laser resurfacing (Experimental): Half of each subject's wound will be treated with a fractional CO2 laser.
  Interventions: Device: Lumenis fractional carbon dioxide laser

INTERVENTIONS:
Device: Lumenis fractional carbon dioxide laser — intra-operative laser resurfacing at time of wound closure
  Other Names: Lumenis
  Arms: Laser resurfacing

SUMMARY:
The purpose of this study is to determine if fractional carbon dioxide laser treatment of a fresh wound at the time of surgery, decreases scar formation. Scar revision is commonly done at 6-10 weeks following surgery. Therefore, it may be more beneficial, for both the patient and physician, to perform scar revision at the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing skin cancer surgery
* Will have a straight-line incision
* Fluent in English
* Must reside in the Los Angeles vicinity for the duration of the study

Exclusion Criteria:

* Non-English speakers
* Pregnant or cognitively impaired subjects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-10; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of scar improvement as assessed by blinded-observer and patient ratings. | At two and six weeks following the procedure

CONTACTS AND LOCATIONS:
Overall Officials: David Ozog, MD, Principal Investigator — Moy-Fincher Medical Group
Locations (1):
- Moy-Fincher Medical Group, Los Angeles, California, United States